CLINICAL TRIAL: NCT02610699
Title: CellScope Oto - Community Pediatric Acceptability Study (CPAS)
Brief Title: Community Pediatric Acceptability Study (CPAS)
Acronym: CPAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other); Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Andi L. Shane, MD, Associate Professor of Pediatrics, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00074526
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Otitis
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smartphone otoscope/Conventional otoscope (Active Comparator): Participating clinicians will use a smartphone otoscope for one month followed by a conventional otoscope for one month, alternating monthly, for a total of 6 months to examine children between 6 months and 18 years of age who have clinical signs of acute otitis media (AOM).
  Interventions: Other: Conventional otoscope; Other: Smartphone otoscope
- Conventional otoscope/Smartphone otoscope (Active Comparator): Participating clinicians will use a conventional otoscope for one month followed by a smartphone otoscope for one month, alternating monthly, for a total of 6 months to examine children between 6 months and 18 years of age who have clinical signs of acute otitis media (AOM).
  Interventions: Other: Conventional otoscope; Other: Smartphone otoscope

INTERVENTIONS:
Other: Conventional otoscope — The conventional analogue otoscope will be used to provide a two-dimensional view of the ear canal. Clinicians will use this for one month periods for a total of 3 months.
Other: Smartphone otoscope — The smartphone otoscope is a pocket size smartphone attachment that uses technology and light source of a smartphone to capture reproducible images of the middle ear and tympanic membrane. Images and videos can be transmitted via real-time communication software from the device to another smartphone. Clinicians will use this for one month periods for a total of 3 months.
  Other Names: CellScope-Oto

SUMMARY:
Ear infections, or otitis media, are a leading cause of health expenditures and antimicrobial prescriptions in children. Diagnosis of otitis media requires the ability to view the tympanic membrane. An instrument called an otoscope with a light source and a magnifying lens with a plastic tip that conforms to the ear canal is currently the standard of care for examining the tympanic membrane. Interpretation of otoscopic examinations is operator-dependent and cannot be seen by anyone other than the person holding the otoscope. A pocket size attachment that uses the technology and light source of a smartphone to capture images of the ear canal and tympanic membrane facilitates image documentation of the otic examination. In previous studies with the device, the investigators have shown that image quality of photographs of the tympanic membrane taken with the smartphone otoscope are equivalent to those taken with a camera-fitted conventional otoscope.

In this study, the Community Provider Assessment Study (CPAS), the investigators will perform a cross-sectional study in which they will randomly assign 3-4 pediatricians to use a smartphone otoscope as the standard of care device for all ear examinations and 3-4 pediatricians to use a conventional otoscope for alternating 1 month periods for 6 months. The parents of children examined during the study period with both devices will be invited to participate in 3 telephone surveys assessing parental satisfaction with the device and antimicrobial use by their child for the otic complaint. The results of this study have the potential to improve diagnosis and management of otitis media, thus improving patient care, reducing costs, and decreasing the opportunity for the development of antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of an otic complaint
* Willing to undergo otoscopy

Exclusion Criteria:

* Unwilling or unable to to complete study telephone questionnaires
* Do not meet inclusion criteria

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Rate of antibiotic prescription following otic examination with smartphone otoscope device compared to conventional otoscope device | 4 weeks following enrollment
  The rate of antibiotic prescription will be assessed by a parent questionnaire. Parents will be asked if they felt comfortable watching and waiting before filling their child's antibiotic prescription. The number of prescriptions filled will be noted.

SECONDARY OUTCOMES:
Time of antibiotic filling following otic examination with smartphone otoscope device compared to conventional otoscope device smartphone otoscope device compared to conventional otoscope device | 4 weeks following enrollment
  The time of filling of the antibiotic prescription will be assessed by a parent questionnaire. Parents will be asked how long they waited before they filled their child's prescription and the response recorded.
Rate of completion of antibiotic course following otic examination with smartphone otoscope device compared to conventional otoscope device | 4 weeks following enrollment
  The rate of completion of the course of antibiotics will be assessed by a parent questionnaire. Parents will be asked if their child completed the course of prescribed antibiotics. The number of children who completed the entire course of antibiotics will be recorded.
Acceptability of management plan following examination with smartphone otoscope device compared to conventional otoscope device | 4 weeks following enrollment
  The acceptability of the management plan following examination with the smartphone otoscope as compared to conventional otoscope will be assessed by a parent questionnaire. A 'yes' response to questions relating to smartphone device images will indicate acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Shane, MD, MPH, MSc, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States